CLINICAL TRIAL: NCT06119815
Title: co2 Gap Changes Versus Inferior Vena Cava Collapsibility in Relation to Cardiac Index as a Prognostic Value in Septic Shock
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Islam Ahmed Ragab, assistant lecturer of anaesthia an icu and pain managment, Sohag University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: soh-Med-23-10-03MD
Record Dates: First submitted 2023-11-01; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: CO2 GAP — CO2 gap will be measured by insertion of radial arterial cannula and internal jugular C.V.P
  * I.V.C collapsibility will be measured by abdominal us at the subcostal area and the IVC diameters will be measured in M-mode coupled to 2D mode 3 cm before the IVC joined the right atrium to ensure that IVC diameter measurements are accurate and that the inter- and intra-observer variability of IVC can be minimized. The IVC collapsibility index (IVCCI) will be calculated as follows: (maximum diameter on expiration (IVC max) - minimum diameter on inspiration (IVC min).
  * Echocardiography for all patients to asses cardiac index in a parasternal (2D) view. The aortic diameter (AoD) will be measured at the aortic valve annulus. The aortic area (AA) will be calculated using the formula: AA = π × (AoD2/ 4). We measured the aortic blood flow using pulsed
  Other Names: IVC collapsibility; echocardiology

SUMMARY:
In 2016, sepsis and septic shock was redocumented as fatal organ dysfunction caused by infection-induced host response disorders (Singer et al. 2016). Infectious shock is a subtype of sepsis; its circulation abnormalities significantly increase the mortality rate. The definition was updated to facilitate rapid identification and timely treatment. Despite the continuous progress of awareness and intervention, the mortality rate of septic shock is approaching 40% or more (Gasim et al. 2016, Karampela et al. 2022).

Infectious shock exists in the presence of imbalance of oxygen supply and demand as well as tissue hypoxia, early improvement of tissue hypoperfusion is key to the treatment, a specific cluster treatment program was recommended in the guidelines of sepsis rescue action (Rhodes et al. 2017).

Severe sepsis remains associated with high mortality, and the early recognition of the signs of tissue hypoperfusion is crucial in its management. The effectiveness of oxygen-derived parameters as resuscitation goals has been questioned, and the latest data have failed to demonstrate clinical advantage (Rudd et al. 2020).

Prompt diagnosis and appropriate treatment of sepsis are of ulmost importance and key to survival. However, routinely used biomarkers, such as C-reactive protein and procalcitonin, have shown moderate diagnostic and prognostic value. Of note, the recent consensus definition for sepsis is based on clinical criteria, implying the paucity of reliable sepsis biomarkers. The new diagnostic criteria also incorporate the use of the SOFA score, a composite prediction tool, which is derived by a combination of clinical signs and biomarkers of organ dysfunction, leaving aside classic inflammatory biomarkers (Pierrakos et al. 2020, Karampela et al. 2022).

The venous oxygen saturation (SvO2) is <70% in the majority of patients with severe sepsis on admission to the intensive care unit (ICU). The central venous-to-arterial carbon dioxide difference or only carbon dioxide gap (PCO2 gap) has gained relevance as a measure of assessment of several parameters (Mallat et al. 2015). The balance of dioxide carbon (CO2) production by the tissues and its elimination through the lungs can be reflected by the difference between the mixed venous content (CvCO2) and the arterial content (CaCO2). This venous-arterial difference in CO2 content (CCO2) can be estimated by the following equation: ΔPCO2 = PvCO2 - PaCO2, denominated PCO2 gap and in physiological conditions it ranges from 2 to 5 mmHg. In a few words, it indicates the difference between partial pressure of carbon dioxide in central venous blood (PvCO2) and arterial blood (PaCO2) (Janotka et al. 2021). The venous-to-arterial carbon dioxide difference (Pv-aCO2) can indicate the adequacy of microvascular blood flow in the early phases of resuscitation in sepsis (Ospina-Tascon et al. 2016, de Sá 2022).

Hence, other resuscitation goals, such as PCO2 gap, have been suggested, due to their ability to predict adverse clinical outcomes and simplicity in patients achieving normal oxygen derived parameters during the early phases of resuscitation in septic shock. The PCO2 gap can be a marker of cardiac output adequacy in global metabolic conditions that are less affected by the impairment of oxygen extraction capacity (Bitar et al. 2020).

ELIGIBILITY:
Inclusion Criteria:

* o Patients with a diagnosis of severe septic shock.

  * Patients With an ICU stay of more than 24 hours

Exclusion Criteria:

* o Age <18 years old.

  * Patients with (COPD).
  * Patients with heart failure.
  * Patients with active pulmonary edema

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-10-10 (Actual); Primary Completion 2025-10-10 (Estimated); Study Completion 2025-10-10 (Estimated)

PRIMARY OUTCOMES:
co2 Gap changes | 24 months
  CO2 gap will be measured by insertion of radial arterial cannula and internal jugular C.V.P 2
IVC collapsibility | 24 months
  I.V.C collapsibility will be measured by abdominal us at the subcostal area and the IVC diameters will be measured in M-mode coupled to 2D mode 3 cm before the IVC joined the right atrium to ensure that IVC diameter measurements are accurate and that the inter- and intra-observer variability of IVC can be minimized. The IVC collapsibility index (IVCCI) will be calculated as follows: (maximum diameter on expiration (IVC max) - minimum diameter on inspiration (IVC min).

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University hospitals, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bakker J, Vincent JL, Gris P, Leon M, Coffernils M, Kahn RJ. Veno-arterial carbon dioxide gradient in human septic shock. Chest. 1992 Feb;101(2):509-15. doi: 10.1378/chest.101.2.509. PMID 1735281
- [Background] Bitar ZI, Maadarani OS, El-Shably AM, Elshabasy RD, Zaalouk TM. The Forgotten Hemodynamic (PCO2 Gap) in Severe Sepsis. Crit Care Res Pract. 2020 Jan 7;2020:9281623. doi: 10.1155/2020/9281623. eCollection 2020. PMID 32377433
- [Background] Blanco P, Aguiar FM, Blaivas M. Rapid Ultrasound in Shock (RUSH) Velocity-Time Integral: A Proposal to Expand the RUSH Protocol. J Ultrasound Med. 2015 Sep;34(9):1691-700. doi: 10.7863/ultra.15.14.08059. Epub 2015 Aug 17. PMID 26283755
- [Background] Bone RC, Balk RA, Cerra FB, Dellinger RP, Fein AM, Knaus WA, Schein RM, Sibbald WJ. Definitions for sepsis and organ failure and guidelines for the use of innovative therapies in sepsis. The ACCP/SCCM Consensus Conference Committee. American College of Chest Physicians/Society of Critical Care Medicine. Chest. 1992 Jun;101(6):1644-55. doi: 10.1378/chest.101.6.1644. PMID 1303622